CLINICAL TRIAL: NCT02604511
Title: Phase II Study of Ibrutinib in Patients With Symptomatic, Previously Untreated Waldenstrom's Macroglobulinemia, and Impact on Tumor Genomic Evolution Using Whole Genome Sequencing
Brief Title: Study of Ibrutinib in Patients With Symptomatic, Previously Untreated Waldenstrom's Macroglobulinemia, and Impact on Tumor Genomic Evolution Using Whole Genome Sequencing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Principal Investigator, Steven Treon, MD, PhD, Steven P. Treon, MD, PhD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-359
Record Dates: First submitted 2015-11-11; First posted 2015-11-13 (Estimated); Results first posted 2022-01-12 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Waldenstrom's Macroglobulinemia
Keywords: Waldenstrom's Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ibrutinib (Experimental): This is single arm, open label, Phase II, single center study designed to evaluate the safety and efficacy of ibrutinib in previously untreated WM patients. Treatment will be administered in 4-week cycles, and participants will receive treatment for up to 48 cycles. Treatment will be comprised of ibrutinib at 420 mg per day by oral administration.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib
  Other Names: Imbruvica; PCI-32765

SUMMARY:
This research study is studying a drug called ibrutinib as a possible treatment for untreated Waldenstrom's Macroglobulinemia (WM).

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has approved ibrutinib as a form of treatment for the patient specific disease.

Ibrutinib has been under investigation in research studies in participants with recurrent B-cell lymphoma, chronic lymphocytic leukemia (CLL), small lymphocytic lymphoma (SLL), mantle cell lymphoma (MCL), diffuse large B-cell lymphoma (DLBCL), and prolymphocytic leukemia, and WM. In a study of ibrutinib in relapsed/refractory WM patients, response rates were high and the treatment was well tolerated.

The prior studies suggest that ibrutinib may be a useful treatment strategy for untreated WM patients. This study will test the safety and efficacy of ibrutinib as an option for untreated WM patients. The study will also conduct genomic sequencing of malignant WM cells before the start of treatment, and 6, 12, 24, 36 and 48 months afterwards. Genomic sequencing is the analysis of the entire DNA structure from tumor and normal cells. The purpose of this sequencing is to study which genetic changes effect how ibrutinib works. The results of these studies could also help in better understanding the course of WM disease, and be applicable to the development of other effective drug treatments.

ELIGIBILITY:
Inclusion Criteria:

* Clinicopathological diagnosis of Waldenstrom's Macroglobulinemia and meeting criteria for treatment using consensus panel criteria from the Second International Workshop on Waldenstrom's macroglobulinemia (Kyle et al, 2003).
* Measurable disease, defined as presence of serum immunoglobulin M (IgM) with a minimum IgM level of ≥ 2 times the upper limit of normal is required.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (see Appendix A.).
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1,000/μL
  * Platelets ≥ 50,000/μL
  * Hemoglobin ≥ 8 g/dL
  * Total bilirubin ≤ 2.0. mg/dL or < 2.5 mg/dL if attributable to hepatic infiltration by neoplastic disease or Gilbert's syndrome.
  * Aspartate aminotransferase (AST or SGOT) and Alanine aminotransferase (ALT or SGPT) ≤ 2.5 X institutional upper limit of normal
  * Estimated Creatinine Clearance ≥30ml/min
* Not on any active therapy for other malignancies with the exception of topical therapies for basal cell or squamous cell cancers of the skin.
* Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or have or will have complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) while participating in the study; and 2) for at least 28 days after discontinuation from the study. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. FCBP must be referred to a qualified provider of contraceptive methods if needed.
* Able to adhere to the study visit schedule and other protocol requirements.
* Ability to understand and the willingness to sign a written informed consent document.
* Both men and women of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

* Prior systemic therapy for WM
* Any serious medical condition, laboratory abnormality, uncontrolled intercurrent illness, or psychiatric illness/social condition that would prevent the participant from signing the informed consent form.
* Concurrent use of any other anti-cancer treatments or any other investigational agents.
* Concomitant use of warfarin or other Vitamin K antagonists.
* Concomitant treatment with strong CYP3A4/5 inhibitor.
* Any condition, including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion could interfere with the absorption or metabolism of ibrutinib.
* Known Central nervous system (CNS) lymphoma.
* Concomitant use of medication known to cause QT prolongation.
* Currently active, clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification, or history of myocardial infarction, unstable angina or acute coronary syndrome within 6 months of screening.
* Malabsorption, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
* Known history of Human Immunodeficiency Virus (HIV), active infection with Hepatitis B Virus (HBV), and/or Hepatitis C Virus (HCV). Subjects who are positive for hepatitis B core antibody or hepatitis B surface antigen must have a negative polymerase chain reaction (PCR) result before enrollment. Those who are PCR positive will be excluded.
* Lactating or pregnant women.
* Inability to swallow capsules.
* History of non-compliance to medical regimens.
* Unwilling or unable to comply with the protocol.
* Major surgery within 4 weeks of first dose of study drug.
* No active infections requiring systemic therapy.
* Known bleeding disorders with the exception of acquired Von Willebrand Disorder suspected on the basis of WM.
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Treon, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massacusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Guijosa A, Ramirez-Gamero A, Sarosiek S, Branagan AR, von Keudell G, Treon SP, Castillo JJ. Ibrutinib plus rituximab vs ibrutinib monotherapy in patients with Waldenstrom macroglobulinemia: a pooled analysis. Blood Adv. 2025 Sep 23;9(18):4705-4715. doi: 10.1182/bloodadvances.2025016536. PMID 40674744
- [Derived] Castillo JJ, Meid K, Gustine JN, Leventoff C, White T, Flynn CA, Sarosiek S, Demos MG, Guerrera ML, Kofides A, Liu X, Munshi M, Tsakmaklis N, Xu L, Yang G, Branagan AR, O'Donnell E, Raje N, Yee AJ, Patterson CJ, Hunter ZR, Treon SP. Long-term follow-up of ibrutinib monotherapy in treatment-naive patients with Waldenstrom macroglobulinemia. Leukemia. 2022 Feb;36(2):532-539. doi: 10.1038/s41375-021-01417-9. Epub 2021 Sep 16. PMID 34531537
- [Derived] Treon SP, Gustine J, Meid K, Yang G, Xu L, Liu X, Demos M, Kofides A, Tsakmaklis N, Chen JG, Munshi M, Chan G, Dubeau T, Raje N, Yee A, O'Donnell E, Hunter ZR, Castillo JJ. Ibrutinib Monotherapy in Symptomatic, Treatment-Naive Patients With Waldenstrom Macroglobulinemia. J Clin Oncol. 2018 Sep 20;36(27):2755-2761. doi: 10.1200/JCO.2018.78.6426. Epub 2018 Jul 25. PMID 30044692

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibrutinib: This is single arm, open label, Phase II, single center study designed to evaluate the safety and efficacy of ibrutinib in previously untreated Waldenstrom's macroglobulinemia (WM) patients. Treatment will be administered in 4-week cycles, and participants will receive treatment for up to 48 cycles. Treatment will be comprised of ibrutinib at 420 mg per day by oral administration.
  Ibrutinib
Period: Overall Study
Arm/Group | Ibrutinib
Started | 31
Completed | 19
Not Completed | 12
Not completed — Adverse Event | 3
Not completed — Disease Progression | 4
Not completed — Withdrawal by Subject | 3
Not completed — Participant ineligible | 1
Not completed — Intercurrent illness | 1

BASELINE CHARACTERISTICS:
Groups:
- Ibrutinib: This is single arm, open label, Phase II, single center study designed to evaluate the safety and efficacy of ibrutinib in previously untreated WM patients. Treatment will be administered in 4-week cycles, and participants will receive treatment for up to 48 cycles. Treatment will be comprised of ibrutinib at 420 mg per day by oral administration.
  Ibrutinib
Arm/Group | Ibrutinib
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 20
Age, Continuous [Median (Full Range); unit: years] | 67 [43 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 28
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Major Response Rate
Description: To asses the percentage of participants with a Partial Response (PR) (50% reduction or more in serum IgM) or better.
Time Frame: 4 years
Population: All participants except one participant determined to be ineligible
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib
Number analyzed (Participants) | 30
Participants | 26

2. Primary Outcome: Best Overall Response Rate
Description: To asses the percentage of participants with an Minor Response (MR) (25% reduction or more in serum IgM) or better.
Time Frame: 4 years
Population: All participants except one participant determined to be ineligible
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib
Number analyzed (Participants) | 30
Participants | 30

3. Secondary Outcome: Duration of Response
Description: The amount of time between attainment of at least a minor response and disease progression.
Time Frame: 6 years
Population: All participants except one determined to be ineligible
Measure: Median (Full Range); unit: months
Groups:
- Ibrutinib: This is single arm, open label, Phase II, single center study designed to evaluate the safety and efficacy of ibrutinib in previously untreated Waldenstrom's macroglobulinemia (WM) patients. Treatment will be administered in 4-week cycles, and participants will receive treatment for up to 48 cycles. Treatment will be comprised of ibrutinib at 420 mg per day by oral administration.
Arm/Group | Ibrutinib
Number analyzed (Participants) | 30
months | 46 [1 to 55]

4. Other Pre Specified Outcome: Time to Response
Description: The amount of time between starting treatment and attaining at least a minor response to therapy
Time Frame: 4 years
Population: All participants except one determined to be ineligible
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ibrutinib
Number analyzed (Participants) | 30
months | 0.9 [0.9 to 1.7]

5. Other Pre Specified Outcome: Progression Free Survival
Description: The number of participants who have not experienced disease progression 6 years after therapy initiation
Time Frame: 6 years
Population: All participants except for one determined to be ineligible
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib
Number analyzed (Participants) | 30
Participants | 24

6. Other Pre Specified Outcome: Overall Survival
Description: The number of participants who are still living 6 years after initiation of ibrutinib
Time Frame: 6 years
Population: All participants except one who was determined to be ineligible
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib
Number analyzed (Participants) | 30
Participants | 30

ADVERSE EVENTS:
Time Frame: Adverse events were collected after ibrutinib initiation, through 30 days of last dose of ibrutinib (e.g. 49 months maximum). Deaths were assessed for up to 6 years.
Arm/Group | Ibrutinib
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 15/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib (N=31)
Head trauma (Injury, poisoning and procedural complications) | 1 (1)
Mania (Psychiatric disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Non-Cardiac Chest pain (General disorders) | 1 (1)
Kidney infection (Renal and urinary disorders) | 1 (1)
Fever (General disorders) | 1 (1)
AST elevation (Investigations) | 2 (2)
ALT elevation (Investigations) | 2 (2)
Drug-induced hepatitis (General disorders) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 1 (1)
Colitis (Infections and infestations) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Esophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Kidney dysfunction (Renal and urinary disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Prostatitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib (N=31)
Anemia (Blood and lymphatic system disorders) | 7 (7)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Ecchymosis (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 5 (5)
Bradycardia (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 5 (5)
Pericarditis (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1)
Blurred vision (Eye disorders) | 3 (3)
Cataract (Eye disorders) | 2 (2)
Conjunctivitis (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 3 (3)
Eye pain (Eye disorders) | 1 (1)
Floaters (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 24 (24)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 5 (5)
Eructation (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 8 (8)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Melena (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 11 (11)
Nausea (Gastrointestinal disorders) | 11 (11)
Oral hemorrhage (Gastrointestinal disorders) | 3 (3)
Oral pain (Gastrointestinal disorders) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
Stomach flu (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 7 (7)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Blood blister (General disorders) | 1 (1)
Brain bleed (General disorders) | 1 (1)
Chills (General disorders) | 10 (10)
Dental implant (General disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 9 (9)
Esophageal spasm (General disorders) | 1 (1)
Fatigue (General disorders) | 22 (22)
Fever (General disorders) | 7 (7)
Flu-like symptoms (General disorders) | 3 (3)
Hernia (General disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 4 (4)
Poison ivy (General disorders) | 1 (1)
Sunburn (General disorders) | 1 (1)
Teeth grinding (General disorders) | 1 (1)
Varicose veins (General disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Bronchial infection (Infections and infestations) | 3 (3)
Herpes zoster (Infections and infestations) | 4 (4)
Influenza (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Lyme disease (Infections and infestations) | 2 (2)
Mucosal infection (Infections and infestations) | 2 (2)
Otitis media (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 2 (2)
Rectum fungus (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 7 (7)
Skin infection (Infections and infestations) | 9 (9)
Soft tissue infection (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 15 (15)
Urinary tract infection (Infections and infestations) | 4 (4)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Bone marrow procedure hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 13 (13)
Calf injury (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 6 (6)
Foot laceration (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Knee injury (Injury, poisoning and procedural complications) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 5 (5)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (3)
Platelet count decreased (Investigations) | 7 (7)
Urine output decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 4 (4)
White blood cell decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (4)
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 (2)
Knee joint hyperflexion (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (19)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mucoid cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Sebaceous cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Carpal tunnel (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 5 (5)
Headache (Nervous system disorders) | 10 (10)
Lethargy (Nervous system disorders) | 2 (2)
Memory impairment (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (6)
Presyncope (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Transient ischemic attack (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 3 (3)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3)
Confusion (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 4 (4)
Renal calculi (Renal and urinary disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Bee sting (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Eczematous Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 8 (8)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 5 (5)
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 (2)
Onychoschizia (Skin and subcutaneous tissue disorders) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (5)
Rash not otherwise specified (Skin and subcutaneous tissue disorders) | 9 (9)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1)
Seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Sensitive skin (Skin and subcutaneous tissue disorders) | 2 (2)
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Skin bleeding (Skin and subcutaneous tissue disorders) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Wart (Skin and subcutaneous tissue disorders) | 1 (1)
Hematoma (Vascular disorders) | 8 (8)
Hypertension (Vascular disorders) | 6 (6)
Phlebitis (Vascular disorders) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT02604511/Prot_SAP_000.pdf